CLINICAL TRIAL: NCT01935973
Title: A Randomized Phase I Study With a Safety Lead-In to Assess the Antitumor Efficacy of the MEK Inhibitor Trametinib Alone or in Combination With GSK2141795, an AKT Inhibitor, in Patients With Recurrent or Persistent Endometrial Cancer NCT #01935973
Brief Title: Trametinib With or Without GSK2141795 in Treating Patients With Recurrent or Persistent Endometrial Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-01659; NCI-2013-01659 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0229O; GOG-0229O (Other: NRG Oncology); GOG-0229O (Other: CTEP); P50CA098258 (NIH); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2013-09-03; First posted 2013-09-05 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Endometrial Adenocarcinoma; Endometrial Clear Cell Adenocarcinoma; Endometrial Mixed Cell Adenocarcinoma; Endometrial Serous Adenocarcinoma; Endometrial Undifferentiated Carcinoma; Recurrent Uterine Corpus Cancer
MeSH Terms: interventions — trametinib; GSK2141795

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (trametinib) (Active Comparator): Patients receive trametinib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving disease progression may cross over to Arm II.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Trametinib
- Arm II (trametinib and Akt inhibitor GSK2141795) (Experimental): Patients receive trametinib PO QD and Akt inhibitor GSK2141795 PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Trametinib; Drug: Uprosertib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Trametinib — Given PO
  Other Names: GSK1120212; JTP-74057; MEK Inhibitor GSK1120212; Mekinist
Drug: Uprosertib — Given PO
  Other Names: GSK2141795; Oral Akt Inhibitor GSK2141795
  Arms: Arm II (trametinib and Akt inhibitor GSK2141795)

SUMMARY:
This randomized phase I trial studies how well trametinib with or without GSK 2141795 (protein kinase B [Akt] inhibitor GSK2141795) works in treating patients with endometrial cancer that has come back (recurrent) or does not go to remission despite treatment (persistent). Trametinib and Akt inhibitor GSK2141795 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether trametinib is a more effective treatment for endometrial cancer when given with or without ATK inhibitor GSK2141795.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the relative activity of trametinib (mitogen-activated protein kinase [MEK] inhibitor) alone or in combination with GSK2141795 (AKT inhibitor) for patients with recurrent or persistent endometrial cancer by progression-free survival. (Phase II) II. To determine the frequency and severity of adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE). (Phase II) III. To determine the tolerability of the combination regimen of trametinib and GSK2141795 through determination of dose-limiting toxicity in a two-stage safety lead in study. (Safety assessment lead-in)

SECONDARY OBJECTIVES:

I. To estimate the association between baseline Kirsten rat sarcoma viral oncogene homolog (KRAS) status and clinical activity (e.g. response and progression-free survival [PFS]) for patients with recurrent or persistent endometrial cancer who are treated with trametinib alone or in combination with GSK2141795.

II. To estimate overall survival (OS) of patients with recurrent or persistent endometrial cancer treated with trametinib therapy alone (excluding patients who cross-over) and trametinib/GSK2141795 combination therapy in the two subgroups of patients defined above.

III. Prognostic factors will be examined for associations with patients who do not crossover.

IV. To estimate objective response and response duration associated with trametinib therapy and trametinib/GSK2141795 combination therapy in the two subgroups of patients defined above.

V. To estimate the relative proportion of patients responding or have 6-month PFS on the therapies administered on this study with those studies that may serve as a historical control.

TERTIARY OBJECTIVES:

I. To estimate the association between baseline genomic biomarkers in the phosphatidylinositol 3 kinase (PI3K)/AKT pathway and clinical activity (e.g. response and PFS) in two subgroups of patients defined above with recurrent or persistent endometrial cancer who are treated with trametinib alone or in combination with GSK2141795.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive trametinib orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving disease progression may cross over to Arm II.

ARM II: Patients receive trametinib PO QD and Akt inhibitor GSK2141795 PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent endometrial carcinoma, which is refractory to curative therapy or established treatments; histologic confirmation of the original primary tumor is required

  * Patients with the following histologic epithelial cell types are eligible: endometrioid adenocarcinoma, serous adenocarcinoma, undifferentiated carcinoma, mixed epithelial carcinoma, uterine clear cell carcinoma, and adenocarcinoma not otherwise specified (N.O.S.)
* Formalin-fixed, paraffin-embedded tumor tissue must be submitted to Baylor College of Medicine (BCM) - Cancer Genetics Laboratory for Clinical Laboratory Improvement Amendments (CLIA)-certified KRAS mutation testing; results must be reported on the eligibility checklist during registration in order to receive treatment assignment

  * Note: if CLIA-certified KRAS mutation tumor testing is available from local or other source (e.g., Foundation Medicine) this report can be submitted to Statistical and Data Center (SDC) to meet this requirement
* All patients must have measurable disease; measurable disease is defined by Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1); measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST version 1.1; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Gynecologic Oncology Group (GOG) performance status of 0 or 1
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy
* Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
* Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration
* Any other prior therapy directed at the malignant tumor, including chemotherapy and immunotherapy, must be discontinued at least three weeks prior to registration; any investigational agent must be discontinued at least 30 days prior to registration
* Any prior radiation therapy must be discontinued at least four weeks prior to registration
* At least 4 weeks must have elapsed since the patient underwent any major surgery (e.g., major: laparotomy, laparoscopy); there is no delay in treatment for minor procedures (e.g., tumor core biopsy)
* Patients must have had one prior chemotherapeutic regimen for management of endometrial carcinoma; initial treatment may include chemotherapy, chemotherapy and radiation therapy, or consolidation/maintenance therapy; chemotherapy administered in conjunction with primary radiation as a radio-sensitizer WILL be counted as a systemic chemotherapy regimen
* Patients are allowed to receive, but are not required to receive, one additional cytotoxic regimen for management of recurrent or persistent disease
* Patients MAY HAVE received non-cytotoxic (biologic or targeted) agent(s) as part of initial treatment and/or for management of recurrent or persistent disease, with the below stated exceptions (see NOTE below); prior hormonal therapy is allowed, but must be discontinued at least one week prior to registration

  * NOTE: Prior therapy with PI3K inhibitors, AKT inhibitors and/or mammalian target of rapamycin (mTor) inhibitors (e.g., everolimus, temsirolimus) is NOT allowed; prior therapy with MEK inhibitors (e.g., AZD6244 or selumetinib) is NOT allowed
* Absolute neutrophil count (ANC) >= 1,500/mcl
* Platelets >= 100,000/mcl
* Hemoglobin >= 9 g/dl
* Creatinine =< 1.5 x institutional/laboratory upper limit of normal (ULN) OR calculated creatinine clearance (Cockcroft-Gault formula) >= 50 ml/min OR 24-hour urine creatinine clearance >= 50 ml/min
* Bilirubin =< 1.5 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN
* Alkaline phosphatase =< 2.5 x ULN
* Albumin >= 2.5 g/dL
* Fasting glucose < 160 mg/dL
* Hemoglobin A1C (HbA1C) =< 8 if patient has diabetes
* Thyroid-stimulating hormone (TSH) within institutional/laboratory normal limits
* Left ventricular ejection fraction (LVEF) greater than or equal to institutional/laboratory lower limit of normal (LLN) by echocardiogram (ECHO) or multi gated acquisition scan (MUGA)
* International normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.5 x ULN
* For patients on Coumadin, INR/prothrombin time (PT)/PTT must be > 1.5 ULN
* Hemodynamic parameters:

  * Systolic blood pressure < 140 mmHg
  * Diastolic blood pressure < 90 mmHg
* All prior treatment-related toxicities must be CTCAE v4 grade =< 1 (except alopecia) at the time of randomization
* Patients with abnormal fasting glucose values at screening will be excluded (fasting glucose >= 160); in addition, patients with type 1 diabetes will also be excluded; however, patients with type 2 diabetes will be allowed if diagnosed >= 6 months prior to enrollment, and if presenting with hemoglobin A1C (HbA1C) =< 8% at screening
* Patients must be able to swallow and retain orally-administered medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation AND for 4 months following discontinuation; women of child-bearing potential must have a negative serum pregnancy test within 14 days prior to randomization; should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately
* Patients must meet pre-entry requirements as specified
* Patients must have signed an approved informed consent and authorization permitting release of personal health information

Exclusion Criteria:

* Patients who have had prior therapy with GSK2141795 or any other PI3K/AKT/MTOR pathway inhibitor
* Patients who have prior therapy with trametinib or any other MEK inhibitor
* Patients who have mucinous, squamous, sarcomas, or carcinosarcomas
* Patient with a history of other invasive malignancies, with the exception of non-melanoma skin cancer are excluded if there is any evidence of other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol eligibility
* Patients with symptomatic or untreated leptomeningeal or brain metastasis or spinal cord compression
* Patients with a history of interstitial lung disease or pneumonitis
* Patients with known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the trametinib, GSK2141795 or dimethyl sulfoxide (DMSO)
* Current use of a prohibited medication; the following medications or non-drug therapies are prohibited:

  * Other anti-cancer therapy while on study treatment
  * Concurrent treatment with bisphosphonates is permitted; however, treatment must be initiated prior to the first dose of study therapy; prophylactic use of bisphosphonates in patients without bone disease is not permitted, except for the treatment of osteoporosis
  * The concurrent use of all herbal supplements is prohibited during the study (including, but not limited to, St. John's Wort, kava, ephedra [ma huang], gingko biloba, dehydroepiandrosterone [DHEA], yohimbe, saw palmetto, or ginseng)
* Drugs that potently inhibit cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) should be prohibited or used with caution; drugs which are strong inducers of CYP3A and may result in lower exposures of GSK2141795 should also be prohibited; drugs that are substrates of CYP3A4 or cytochrome P450 family 2, subfamily C, polypeptide 8 (CYP2C8) with a narrow therapeutic index may be prohibited; drugs that are sensitive substrates of CYP3A4 or CYP2C8 should be used with caution

  * Caution should be exercised when dosing trametinib concurrently with medications with narrow therapeutic windows that are substrates of CYP2C8; drugs that potently inhibit or induce CYP3A4 should be administered with caution
  * Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
  * The following medications (including but not limited to) are prohibited during the study:

    * PROHIBITED-highly sensitive and/or low therapeutic index

      * Cisapride
      * Pimozide
      * Astemizole
      * Rosuvastatin, sulfasalazine
    * PROHIBITED-strong inducers/inhibitors of CYP3A4

      * Clarithromycin, telithromycin, rifamycin class agents (e.g., rifampin, rifabutin, rifapentine), troleandomycin
      * Itraconazole, ketoconazole
      * Nefazodone
      * Atazanavir, delavirdine, indinavir, lopinavir, nelfinavir, ritonavir, saquinavir, nevirapine
      * Carbamazepine, phenobarbital, phenytoin
  * The following medications (including but not limited to) that may alter the concentrations of trametinib or GSK2141795 or have their elimination altered by trametinib or GSK2141795 should be administered WITH CAUTION:

    * USE WITH CAUTION-Drugs potentially affecting trametinib or GSK2141795 concentrations

      * Quinidine, diltiazem, verapamil
      * Fluvoxamine, fluoxetine, paroxetine, nefazodone
      * Aprepitant, cimetidine
      * Fluconazole, terbinafine, voriconazole
      * Ciprofloxacin, erythromycin, isoniazid
      * Mibefradil, diltiazem, verapamil
      * Aprepitant, oxandrolone, tizanidine, gemfibrozil
    * USE WITH CAUTION-Drugs that may inhibit permeability (P)-glycoprotein (gp) and breast cancer resistance protein (BCRP)

      * Valspodar
      * Atorvastatin
      * Carvedilol
      * Methadone
      * Meperidine
      * Omeprazole
    * USE WITH CAUTION-Drugs that may have their concentrations altered by trametinib or GSK2141795

      * Repaglinide, rosiglitazone, pioglitazone
      * Alfentanil, fentanyl
      * Quinidine
      * Cilostazol
      * Astemizole
      * Diergotamine, ergotamine, eletriptan
      * Pimozide
      * Buspirone
      * Felodipine
      * Sildenafil, tadalafil, vardenafil
      * Cerivastatin, lovastatin, simvastatin, atorvastatin
      * Alprazolam, diazepam, midazolam, triazolam
      * Cyclosporine, sirolimus, tacrolimus
      * Cisapride
      * Cyclosporine, torsemide, chloroquine, zopiclone
      * Eplerenone
      * Chloroquine, zopiclone
    * Use of repaglinide, rosiglitazone and/or pioglitazone is permitted only after consultation with the Cancer Therapy Evaluation Program (CTEP) Medical Monitor
* Known hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (unless cleared) will be excluded
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* History or current evidence/risk of retinal vein occlusion (RVO)
* History or evidence of cardiovascular risk including any of the following:

  * LVEF < LLN
  * A QT interval corrected for heart rate using the Bazett's formula (QTcB) >= 480 msec
  * History or evidence of current clinically significant uncontrolled arrhythmias (exception: patients with controlled atrial fibrillation for > 30 days prior to registration are eligible)
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to registration
  * History or evidence of current >= class II congestive heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * Treatment-refractory hypertension defined as a blood pressure of systolic > 140 mmHg or diastolic > 90 mmHg which cannot be controlled by anti-hypertensive therapy
  * Patients with intra-cardiac defibrillators or permanent pacemakers
  * Known cardiac metastases
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients who are pregnant or nursing; women of childbearing potential should be advised to avoid pregnancy and use effective methods of contraception; if a patient becomes pregnant while the patient receives trametinib and/or GSK2141795, the potential hazard to the fetus should be explained to the patient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2015-09-08 (Actual); Study Completion 2015-09-08 (Actual)

PRIMARY OUTCOMES:
PFS by regimen administered using RECIST version 1.1 (Phase II) | The duration of time from study entry to time of progression or death, whichever occurs first, assessed up to 5 years
  The null hypothesis will be tested against the alternative with a stratified log-rank test.
Frequency of adverse events defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related | Up to 30 days after last study treatment
  Reported using the descriptions found in the National Cancer Institute (NCI) CTCAE version 4.0.
Severity of adverse events, graded using the NCI CTCAE version 4.0 (Safety assessment and phase II) | Up to 30 days after last study treatment
Incidence of dose-limiting toxicity (DLT), graded according to the current version of NCI CTCAE (Safety assessment) | 28 days
  If 3 or fewer patients out of 12 experience DLTs in course 1 (including treatment delays for course 2 of greater than 2 weeks due to toxicities), then the regimen will be deemed safe for administration in the phase II study. If 4 or more patients out of 12 experience DLTs, then the regimen will be declared unsafe.

SECONDARY OUTCOMES:
KRAS status (mutant or wild type) | Baseline
  The impact of KRAS mutation on response and PFS will be assessed according to the regimens administered. Given the possibility that KRAS+ patients may be small in number (20%), these comparisons may be informal (e.g. Kaplan-Meier survival estimates).
Tumor response by regimen, assessed using RECIST | Up to 5 years
PFS by regimen | The duration of time from study entry to time of progression or death, whichever occurs first, assessed up to 5 years
OS by regimen | The duration of time from study entry to time of death or the date of last contact, assessed up to 5 years
  Overall survival will be compared by regimen with log-rank tests and Cox modeling.
Response duration by KRAS mutation and regimen | From the first date of response until disease progression or death, assessed up to 5 years
  Response duration will be assessed with Kaplan-Meier curves.
Proportion of responding patients | Up to 5 years

OTHER OUTCOMES:
Baseline genomic biomarkers | Baseline
  Baseline genomic biomarkers will be assessed against response, PFS, OS (excluding crossovers) by regimen and KRAS status through odds ratios and proportional hazards estimates where possible.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon N Westin, Principal Investigator — NRG Oncology
Locations (22):
- United States (22):
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Augusta University Medical Center, Augusta, Georgia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - M D Anderson Cancer Center, Houston, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia